CLINICAL TRIAL: NCT04864223
Title: A New Approach to Classifying and Predicting Long-term Bothersome Pain and Functional Decline in Older Adults
Brief Title: Classifying and Predicting Long-term Pain and Function in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sean Rundell, Assistant Professor, University of Washington
Other Study IDs: STUDY00005507
Record Dates: First submitted 2019-08-14; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain; Pain
Keywords: older adults; chronic pain; function; physical performance
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will use novel methods to detect clinically meaningful subgroups of older adults based on long-term trajectories of bothersome pain and function. It will then identify older adults at high risk of experiencing poor long-term pain and function. Anticipated results will provide new insights into long-term patterns of pain and function across the aging process and identify potential predictors of each trajectory.

DETAILED DESCRIPTION:
The long-term goal of this planned line of research is to reduce the burden of pain and maximize function in older adults as they age. This line of research will begin by completing the following Aims: Aim 1) Identify and describe clinically meaningful long-term trajectories of bothersome pain and functional decline in a population-based sample of older adults and Aim 2) Estimate the association between candidate prognostic factors typically available in electronic health records and long-term bothersome pain and function trajectories to inform the development of eventual risk prediction models. This will be a retrospective cohort study using longitudinal data from the population-based National Health and Aging Trends Study (NHATS). This project will use novel methods to identify clinically meaningful subgroups of older adults based on long-term trajectories of bothersome pain and function. Group-based trajectory modeling (GBTM) is a novel method to model dynamic phenomena such as pain and function. Older adults at high risk of experiencing poor long-term pain and function outcomes will be identified by leveraging potential prognostic factors typically available in electronic health records or administrative data. It is anticipated that our results will provide new insights into long-term patterns of pain and function across the aging process and identify potential predictors of each trajectory.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older adults from Round 1 of the NHATS cohort

Exclusion Criteria:

* participants who are non-ambulatory (require a wheelchair or scooter for mobility) at Round 1

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: NHATS is a cohort of older adults and is representative of Medicare beneficiaries age 65 years and older. It is a "unique national resource for the scientific study of functioning in later life." The sample is drawn from the Medicare enrollment files, and the survey oversamples Blacks and those at older ages. NHATS data collection began in 2011 (Round 1) with in-person interviews. Participants were re-interviewed yearly (Rounds 2-7). This is a unique cohort because it contains comprehensive survey data in addition to physical performance measures for individuals over multiple years. During each round, NHATS collects a wide array of information during the interviews, including: demographic, health, social, economic, environmental, cognitive, behavioral, and physical data.
Sampling Method: Probability Sample
Enrollment: 6783 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Bothersome Pain | 6 years
  Question: "In the last month, have you been bothered by pain?" Dichotomous response of yes or no
Physical Performance | 6 years
  Short Physical Performance Battery (SPPB). Scored from 0=worst to 12=best based on 3 performance tests: walking, chairs stands, and balance tasks

SECONDARY OUTCOMES:
Activity Limitations Due to Pain | 6 years
  Question: "In the last month, has pain ever limited your activities?" Dichotomous response of yes or no
Functional Capacity | 6 years
  Self-reported physical capacity. A composite score of self-reported ability to do six pairs of activities: walking 3 or 6 blocks independently, climbing 10 or 20 stairs, lifting and carrying 10 or 20 pounds, bending over or kneeling down, reaching overhead or placing a heavy object overhead, and grasping small objects or opening a jar. Scores range 0-12 with higher scores indicating greater capacity to perform these activities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is publically available at https://www.nhats.org/